CLINICAL TRIAL: NCT06846567
Title: A Phase I Clinical Study Evaluating the Safety, Pharmacokinetics, Food Effect, Single-Dose Proportionality, and Multiple-Dose Pharmacokinetic Comparison With Melogabalin Besilate Tablets After Single and Multiple Oral Administrations of BM2216 Extended-Release Tablets in Healthy Adult Subjects.--Single-Center, Randomized, Open-Label, Parallel/Crossover Design.
Brief Title: Phase I Study of BM2216 ER vs. Melogabalin Besilate: Safety, PK, and Food Effect in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Anglikang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BM-CR-2216-101P/102P/103P
Record Dates: First submitted 2025-02-17; First posted 2025-02-26 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Neuropathies; Diabetes Mellitus
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part 1 (Experimental): BM2216 Extended-Release Tablets（test drug，16.5mg）：one tablet on an empty stomach and one tablet after a meal,Three cycles, take once per cycle； Mirogabalin Besilate Tablets(reference drug,15mg)：Take half a tablet orally once on an empty stomach,Three cycles, take twice per cycle.
  Interventions: Drug: Mirogabalin Besilate Tablets; Drug: BM2216 Extended-Release Tablets(16.5mg)
- Part 2 (Experimental): BM2216 Extended-Release Tablets（test drug，5.5mg、11mg）:one tablet after dinner,Single cycle, take once per cycle; BM2216 Extended-Release Tablets（test drug，16.5mg）：Administer one tablet after dinner (16.5mg dose group); administer two tablets after dinner (33mg dose group)，Single cycle, take once per cycle.
  Interventions: Drug: BM2216 Extended-Release tablets（5.5mg）; Drug: BM2216 Extended-Release Tablets(11mg); Drug: BM2216 Extended-Release Tablets(16.5mg)
- Part 3 (Experimental): BM2216 Extended-Release Tablets(test drug,16.5mg)：Administer one tablet after dinner.Bicyclic, with continuous administration for 4 days each cycle.
  Mirogabalin Besilate Tablets(reference drug,15mg)：Take half a tablet orally once on an empty stomach，Two cycles, administer continuously for 4 days per cycle (take 8 times per cycle).
  Interventions: Drug: Mirogabalin Besilate Tablets; Drug: BM2216 Extended-Release Tablets(16.5mg)

INTERVENTIONS:
Drug: BM2216 Extended-Release tablets（5.5mg） — 5.5mg BM2216 Extended-Release ,test drug
  Arms: Part 2
Drug: Mirogabalin Besilate Tablets — 15mg of Mirogabalin Besilate Tablets,reference drug
  Arms: Part 1; Part 3
Drug: BM2216 Extended-Release Tablets(11mg) — 11mg of BM2216 Extended-Release,test drug
  Arms: Part 2
Drug: BM2216 Extended-Release Tablets(16.5mg) — 16.5mg of BM2216 Extended-Release Tablets,test drug

SUMMARY:
A Phase I Clinical Study Evaluating the Safety, Pharmacokinetics, Food Effect, Single-Dose Proportionality, and Multiple-Dose Pharmacokinetic Comparison with Melogabalin Besilate Tablets after Single and Multiple Oral Administrations of BM2216 Extended-Release Tablets in Healthy Adult Subjects. To evaluate the pharmacokinetic characteristics of BM2216 Extended-Release Tablets in healthy adult subjects under fasting and postprandial conditions, and to assess the impact of food; to evaluate the dose proportionality following a single administration.To compare the single and multiple dose pharmacokinetic characteristics of BM2216 Extended-Release Tablets with those of Melogabalin Besilate Tablets, and to determine the relative bioavailability.To assess the safety of BM2216 Extended-Release Tablets in healthy adult subjects following single and multiple oral administrations.

DETAILED DESCRIPTION:
This study is divided into three parts: PART-1, PART-2, and PART-3. It is planned that PART-2 will prioritize enrollment (all dose groups can be enrolled simultaneously), while PART-1 and PART-3 can also be enrolled concurrently. The doses for PART-1 and PART-3 may be adjusted based on the results of PART-2.

PART-1 (FE + Single-Dose PK Comparison):

A Single-Center, Randomized, Open-Label, Three-Period, Three-Sequence, Three-Way Crossover Study to Evaluate the Pharmacokinetic Characteristics and Food Effect of BM2216 Extended-Release Tablets After Single Oral Administration Under Fasting and High-Fat Meal Conditions in Healthy Adult Subjects, and to Compare the Pharmacokinetic Characteristics with Multiple-Dose Melogabalin Besilate Tablets, Relative Bioavailability, and Safety. This study plans to enroll 18 subjects, who will be randomly assigned to three dosing sequence groups in a 1:1:1 ratio.

PART-2 (Single-Dose Proportionality):

A single-center, open-label, parallel design will be used to evaluate the pharmacokinetic characteristics, dose proportionality, and safety of BM2216 extended-release tablets after a single dose in healthy adult subjects. This study plans to enroll 32 subjects, with four dose groups of BM2216 extended-release tablets (5.5 mg, 11 mg, 16.5 mg, and 33 mg), with 8 subjects in each group.

PART-3 (Multiple-Dose PK Comparison):

This study adopts a single-center, randomized, open-label, two-period, two-sequence, two-crossover design to evaluate the pharmacokinetic characteristics of BM2216 extended-release tablets after multiple oral doses in healthy adult subjects, as well as the pharmacokinetic comparison with multiple doses of mirogabalin besylate tablets, relative bioavailability, and safety. The study plans to enroll 16 subjects, who will be randomly assigned to two dosing sequence groups in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before the trial and fully understand the trial content, procedures, and potential adverse reactions;
2. Be able to complete the study in accordance with the trial protocol requirements;
3. The subject (and their partner) is willing to voluntarily adopt effective contraceptive measures from screening until 6 months after the last administration of the study drug. Specific contraceptive measures are detailed in Appendix 3;
4. Male and female subjects aged 18-45 years (inclusive);
5. Male subjects must weigh no less than 50.0 kg, and female subjects must weigh no less than 45.0 kg. BMI = weight (kg) / height (m²), with a body mass index ranging from 19.0 to 26.0 kg/m² (inclusive).

Exclusion Criteria:

1. Average daily smoking of more than 5 cigarettes within the 3 months prior to screening;
2. Allergy to any component of the investigational product, or a history of drug, food, or other substance allergies, or a history of allergic diseases;
3. History of drug abuse and/or alcoholism (alcoholism defined as consuming more than 14 units of alcohol per week: 1 unit = 285 mL of beer, 25 mL of spirits, or 100 mL of wine); history of drug abuse or use of illicit drugs within the past 5 years;
4. Donation of blood or significant blood loss (>450 mL) within the 3 months prior to screening;
5. Difficulty swallowing or a history of gastrointestinal, liver, or kidney diseases (regardless of cure status) or surgeries within the 6 months prior to screening that may affect drug absorption or excretion;
6. Use of strong inhibitors and/or inducers of hepatic metabolic enzymes (CYP1A2, 2B6, 2A6, 2C8, 2C19, 3A4, and 3A5) within 28 days prior to the first dose. Strong inhibitors include ciprofloxacin, clopidogrel, itraconazole, ketoconazole, ritonavir, troleandomycin, etc. Strong inducers include rifampicin, carbamazepine, phenytoin sodium, St. John's wort, etc. Use of inhibitors or inducers of absorption transporters (e.g., P-gp, BCRP, OATP) and efflux transporters within 28 days prior to the first dose. For details, refer to Appendix 4;
7. Use of any prescription drugs, over-the-counter drugs, health supplements, or herbal medicines within 14 days prior to the first dose;
8. Consumption of any caffeine-rich, xanthine-rich, or CYP3A4 metabolism-affecting foods/beverages (e.g., grapefruit, animal liver, coffee, tea, cola, chocolate, etc.) within 14 days prior to the first dose or during the trial, or engagement in strenuous exercise (e.g., strength training, aerobic training, soccer), or other factors that may affect drug absorption, distribution, metabolism, or excretion;
9. Significant changes in diet or exercise habits within 7 days prior to the first dose;
10. Participation in another clinical trial within the 3 months prior to screening (subjects who withdrew from the study before treatment, i.e., were not randomized or did not receive treatment, may be enrolled in this study);
11. Inability to tolerate high-fat meals or having special dietary requirements, and unwillingness to accept a standardized diet;
12. Abnormal vital signs during screening (ear temperature <35.7°C or >37.5°C; pulse <60 bpm or >100 bpm; systolic blood pressure <90 mmHg or ≥140 mmHg, diastolic blood pressure <60 mmHg or ≥90 mmHg);
13. Clinically significant abnormalities in 12-lead electrocardiogram (ECG);
14. Female subjects who are breastfeeding or have a positive pregnancy test during screening or the trial period;
15. Clinically significant abnormalities in clinical laboratory tests or other clinically significant diseases (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, pulmonary, immunological, psychiatric, or cardiovascular diseases) identified prior to screening;
16. Positive screening results for viral hepatitis (including hepatitis B and C), HIV antibodies, or syphilis antibodies;
17. Occurrence of acute illness from the screening phase until before study drug administration;
18. Consumption of any alcohol-containing products within 24 hours prior to the first dose or a positive alcohol breath test;
19. Positive urine drug screening;
20. Inability to tolerate venipuncture or a history of needle or blood phobia;
21. Vaccination within 4 weeks prior to the first dose or planned vaccination during the study period;
22. Other conditions deemed by the investigator to make the subject unsuitable for participation in the clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-01-12 (Actual)

PRIMARY OUTCOMES:
The plasma concentration of study drugs | Blood samples were collected from 0 hours to 32 hours after administration.
  Plasma concentration of study drugs will be measured at all the time points.

SECONDARY OUTCOMES:
Frequency of occurrence of adverse events | 0 hours to 48 hours after administration.
  Any adverse event were classified by severity, treatment and its relationship with the study drug was evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing Bishan People's Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No